CLINICAL TRIAL: NCT00421811
Title: An Open-Label, Multicenter, Phase 1/2 Dose Escalation Study to Evaluate Safety, Tolerability and Anti-tumor Activity of Systemic ADH-1 in Combination With Normothermic Isolated Limb Infusion of Melphalan in Subjects With Locally Advanced In-Transit Malignant Melanoma (Adherex Protocol Number AHX-01-007).
Brief Title: A Study of ADH-1 in Combination With Normothermic Isolated Limb Infusion of Melphalan
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adherex Technologies, Inc. (Industry)
Responsible Party: Clinical Study Manager, Adherex Technologies, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHX-01-007
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Neoplasms
Keywords: cancer; tumors; melanoma; anticarcinogenic agents; antineoplastic agents; cadherins; solid tumors
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — Melphalan

INTERVENTIONS:
Drug: ADH-1 — 4 gm IV Days 1 and 8
Drug: melphalan — By Isolated Limb Infusion (ILI), Lower Extremity: 7.5 mg/L (Limb Volume), Day 1 or Upper Extremity: 10 mg/L (Limb Volume), Day 1

SUMMARY:
N-cadherin, a protein involved in blood vessel cell binding and on the surface of many tumor cells, is increased as cancer progresses. ADH-1 blocks N-cadherin. This study will test the safety and effects of the combination ADH-1 with Normothermic Isolated Limb Infusion of Melphalan in subjects with locally advanced malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male and female patients > or = 18 years of age with diagnosis of melanoma for which treatment with Normothermic Isolated Limb Infusion (ILI) of melphalan would be appropriate
* Measurable disease
* Disease site(s) must be distal to the planned site of tourniquet placement
* Available for immunohistochemical testing of N-cadherin expression tumor tissue
* Adequate performance status and organ function, as evidenced by hematological and biochemical blood testing and ECG

Exclusion Criteria:

* Receipt of ADH-1 prior to this clinical study (prior melphalan via ILI, is okay)
* Stage IV melanoma
* Chemotherapy, radiotherapy, or any other investigational drug within 4 weeks before study entry
* History of tumors that have shown clinically significant evidence of active bleeding within 12 weeks before study entry
* Stroke, major surgery, or other major tissue injury within 4 weeks before study entry
* Uncontrolled congestive heart failure, coronary artery disease, or life threatening arrhythmias; myocardial infarction within 12 months; significant electrocardiogram (ECG) abnormalities
* Allergic reaction to any therapeutic peptide or to melphalan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To tabulate the Best Overall Response according to unconfirmed RECIST, modified for cutaneous lesions | By Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Doug Tyler, MD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - University of Colorado, Denver, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah

REFERENCES:
- See also: (Adherex Technologies Inc. Corporate Homepage) — http://www.adherex.com